CLINICAL TRIAL: NCT03228875
Title: Early Life Origins of Pediatric and Adult Diseases: Boston Birth Cohort Study
Brief Title: Boston Birth Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Boston Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00022869
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Maternal Health; Child Health; Pregnancy Complications; Birth Outcome, Adverse
Keywords: Boston Birth Cohort; Early life origins of pediatric and adult disease; Gene environment interaction; Health across life course and generations
MeSH Terms: conditions — Pregnancy Complications; Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 21 Years
Biospecimen Retention: Samples With DNA — Plasma, red blood cell, placenta, urine, DNA, RNA, Swab, Stool
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Early life exposures may lead to adverse effects on health in later life. The Boston birth Cohort study is designed to study a broad array of early life factors and their effects on maternal and child health outcomes.

DETAILED DESCRIPTION:
Any woman admitted to the Labor and Delivery floor at the Boston Medical Center (BMC) who delivers a singleton live infant and meets our case (gestational age <37 weeks or birthweight <2,500 grams) or control (full term birth with birthweight >2,500 grams) criteria will be eligible.

Postnatal follow-up of enrolled mother-child pair is conducted from birth to age 21 years.

The Boston Birth Cohort has high-quality biospecimen collection, and comprehensive epidemiological, clinical, and environmental exposure data via standardized questionnaire interview, measurements, and review of the electronic medical records.

ELIGIBILITY:
Inclusion Criteria:

* Mothers who deliver singleton live births at Boston Medical Center are eligible for the study.

Exclusion Criteria:

* pregnancies that are a result of in vitro fertilization or that involve multiple gestations, fetal chromosomal abnormalities or major birth defects.

Ages: 0 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: US, predominantly urban, BIPOC (Black, Indigenous, and people of color).
Sampling Method: Non-Probability Sample
Enrollment: 24000 (Estimated)
Dates: Start 1998-10 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Pregnancy complications | At birth
  Multiple pregnancy complications are examined including gestational diabetes, hypertensive disorders of pregnancy.
Birth outcomes - preterm birth | At birth
  Birth outcomes are examined - preterm birth.
Birth outcomes - birthweight | At birth
  Birth outcomes are examined - birthweight.
Child health outcomes | From birth to 21 years
  Multiple child health outcomes are examined including food allergy, asthma, child's overweight or obesity, blood pressure, and child neuro-developmental outcomes.
Maternal health outcomes | After delivery to 21 years
  Multiple maternal health outcomes are measured including blood pressure, weight, height, physician diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Xiaobin Wang, MD, ScD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yaskolka Meir A, Wang G, Hong X, Hu FB, Wang X, Liang L. Newborn DNA methylation age differentiates long-term weight trajectories: the Boston Birth Cohort. BMC Med. 2024 Sep 11;22(1):373. doi: 10.1186/s12916-024-03568-9. PMID 39256781
- [Derived] Cameron K, Borahay M, Hong X, Baker V, Vaught A, Wang X. Uterine fibroids and risk of hypertensive disorders of pregnancy - results from a racially diverse high-risk cohort. medRxiv [Preprint]. 2024 Mar 7:2024.03.05.24303830. doi: 10.1101/2024.03.05.24303830. PMID 38496516
- [Derived] Hong X, Rosenberg AZ, Heymann J, Yoshida T, Waikar SS, Ilori TO, Wang G, Rebuck H, Pearson C, Wang MC, Winkler CA, Kopp JB, Wang X. Joint Associations of Pregnancy Complications and Postpartum Maternal Renal Biomarkers With Severe Cardiovascular Morbidities: A US Racially and Ethnically Diverse Prospective Birth Cohort Study. J Am Heart Assoc. 2023 Nov 21;12(22):e029311. doi: 10.1161/JAHA.122.029311. Epub 2023 Nov 10. PMID 37947096
- [Derived] McArthur KL, Zhang M, Hong X, Wang G, Buckley JP, Wang X, Mueller NT. Trimethylamine N-Oxide and Its Precursors Are Associated with Gestational Diabetes Mellitus and Pre-Eclampsia in the Boston Birth Cohort. Curr Dev Nutr. 2022 Jun 21;6(7):nzac108. doi: 10.1093/cdn/nzac108. eCollection 2022 Jul. PMID 35949367
- [Derived] Huang W, Igusa T, Wang G, Buckley JP, Hong X, Bind E, Steffens A, Mukherjee J, Haltmeier D, Ji Y, Xu R, Hou W, Tina Fan Z, Wang X. In-utero co-exposure to toxic metals and micronutrients on childhood risk of overweight or obesity: new insight on micronutrients counteracting toxic metals. Int J Obes (Lond). 2022 Aug;46(8):1435-1445. doi: 10.1038/s41366-022-01127-x. Epub 2022 May 19. PMID 35589962
- [Derived] Lee ASE, Ji Y, Raghavan R, Wang G, Hong X, Pearson C, Mirolli G, Bind E, Steffens A, Mukherjee J, Haltmeier D, Fan ZT, Wang X. Maternal prenatal selenium levels and child risk of neurodevelopmental disorders: A prospective birth cohort study. Autism Res. 2021 Dec;14(12):2533-2543. doi: 10.1002/aur.2617. Epub 2021 Sep 24. PMID 34558795
- [Derived] Olapeju B, Hong X, Wang G, Summers A, Burd I, Cheng TL, Wang X. Birth outcomes across the spectrum of maternal age: dissecting aging effect versus confounding by social and medical determinants. BMC Pregnancy Childbirth. 2021 Sep 1;21(1):594. doi: 10.1186/s12884-021-04077-w. PMID 34470614
- [Derived] Olapeju B, Ahmed S, Hong X, Wang G, Summers A, Cheng TL, Burd I, Wang X. Maternal Hypertensive Disorders in Pregnancy and Postpartum Plasma B Vitamin and Homocysteine Profiles in a High-Risk Multiethnic U.S., Population. J Womens Health (Larchmt). 2020 Dec;29(12):1520-1529. doi: 10.1089/jwh.2020.8420. Epub 2020 Nov 16. PMID 33252313